CLINICAL TRIAL: NCT03008122
Title: Phase I, Randomized, Double-blinded, Placebo-Controlled Dose De-escalation Study to Evaluate the Safety and Immunogenicity of Alum Adjuvanted Zika Virus Purified Inactivated Vaccine (ZPIV) Administered by the Intramuscular Route in Adult Subjects Who Reside in a Flavivirus Endemic Area
Brief Title: Phase I, Randomized, Double-blinded, Placebo-Controlled Dose De-escalation Study to Evaluate Safety and Immunogenicity of Alum Adjuvanted Zika Virus Purified Inactivated Vaccine (ZPIV) in Adults in a Flavivirus Endemic Area
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-0034; HHSN272201300021I
Record Dates: First submitted 2016-12-15; First posted 2017-01-02 (Estimated); Results first posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2018-01

CONDITIONS: Zika Virus Infection
Keywords: Flavivirus; Inactivated; Phase I; Vaccine; ZIKA; ZPIV
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): 5 mcg ZPIV administered IM in a homologous prime-boost regimen on Day 1 and Day 29 , n=45 (2 sentinels, 43 non-sentinels) or placebo, n=5
  Interventions: Other: Placebo; Biological: Zika Virus Purified Inactivated Vaccine (ZPIV)
- Group 2 (Experimental): 2.5 mcg ZPIV administered IM in a homologous prime-boost regimen on Day 1 and Day 29, n=35 or placebo, n=5
  Interventions: Other: Placebo; Biological: Zika Virus Purified Inactivated Vaccine (ZPIV)

INTERVENTIONS:
Other: Placebo — Placebo
Biological: Zika Virus Purified Inactivated Vaccine (ZPIV) — Zika Virus Purified Inactivated Vaccine with aluminum hydroxide adjuvant.

SUMMARY:
This study is randomized, double-blinded, placebo-controlled, Phase 1, dose de-escalation study to evaluate the safety, reactogenicity, and immunogenicity of Alum Adjuvanted Zika Virus Purified Inactivated Vaccine (ZPIV) administered to healthy male and non-pregnant female adult subjects. This study will enroll 90 healthy male and non-pregnant female subjects between the ages of 21 and 49 and will be conducted at Ponce Medical School Foundation, Inc.-CAIMED in Ponce, Puerto Rico. The duration of each subject's participation is approximately 26 months from recruitment through the last study visit. The entire study is expected to take approximately 49 months to complete. Two dose levels will be evaluated. Each subject will receive either placebo or 5 mcg (Group 1) or 2.5 mcg (Group 2) of ZPIV administered by intramuscular (IM) injection on Days 1 and 29. Solicited local and systemic reactogenicity data will be collected from all subjects through Day 8 after each vaccination. All subjects will be monitored for occurrence of unsolicited adverse events until 28 days after the second vaccination. The study will consist of a screening period of up to 28 days, a vaccination period in which subjects will receive a prime dose of vaccine on Day 1 followed by a boost on Day 29, and a follow-up period of 24 months post boost vaccination. Primary objectives are: 1) Assess the safety and reactogenicity of a homologous prime boost regimen of ZPIV given at two different dose levels. 2) Compare the safety and reactogenicity of ZPIV after each vaccination, between dosage groups, and by pre-vaccination flavivirus immune status.

DETAILED DESCRIPTION:
This study is a single-center, randomized, double-blinded, placebo-controlled, Phase 1, dose de-escalation study to evaluate the safety, reactogenicity, and immunogenicity of a purified inactivated, alum-adjuvanted ZIKV vaccine (ZPIV) administered in a homologous prime-boost regimen to healthy male and non-pregnant female adult subjects living in a flavivirus-endemic area. This study will enroll 90 subjects between the ages of 21 and 49 and will be conducted at Ponce Medical School Foundation, Inc.-CAIMED in Ponce, Puerto Rico. The entire duration of each subject's participation is approximately 26 months including recruitment and collection of data on the safety and reactogenicity of the study vaccine and collection of samples for the assessment of immunogenicity. This study is expected to take approximately 49 months to complete. Two dose levels will be evaluated. Each subject will receive either placebo or 5 mcg (Group 1) or 2.5 mcg (Group 2) of ZPIV administered by intramuscular (IM) injection on Days 1 and 29. The study will consist of a screening period of up to 28 days, a vaccination period in which subjects will receive a prime dose of vaccine on Day 1 followed by a homologous boost on Day 29, and a follow-up period of 24 months post boost vaccination. The study will begin with enrollment of 2 sentinel subjects in Group 1 who will receive 5 mcg ZPIV open label. One sentinel subject will be vaccinated, followed for one day for safety and reactogenicity, and if no halting rules are met per determination of the PI and co-PI, then the second sentinel subject will receive 5 mcg ZPIV open-label. Both sentinels will be followed for safety through Day 8 and if no predefined halting rules are met and no safety concerns are identified, then enrollment of the Group 1 non-sentinel subjects will proceed in double-blind fashion. The same procedure will be used for administration of the boost vaccination to the Group 1 sentinels: 1 sentinel (can be either) will receive 5 mcg ZPIV open-label, be followed for one day for safety and reactogenicity, and if no halting rules are met, then the 2nd sentinel will receive the boost vaccine. Both sentinels will be followed until Day 8 after 2nd vaccination for safety and reactogenicity and if no halting rules are met, then boost vaccination of the Group 1 non-sentinel subjects can proceed. Enrollment of the 2.5 mcg ZPIV group (Group 2) can begin after or at the same time non-sentinel subjects in Group 1 receive the 1st dose of vaccine. As of December 18, 2017, the majority of non-sentinel subjects in Group 1 have already received the 1st dose and have been followed until Day 8 for safety and reactogenicity, and no halting rules have been met or safety concerns identified. As this is a dose de-escalation study, concurrent enrollment of some remaining non-sentinel subjects in Groups 1 is permitted after enrollment of Group 2 subjects has begun; also, no sentinel subjects will be used in Group 2. All subjects in Group 2 will receive study product or placebo in double-blind fashion. The original study design planned to enroll 40 ZPIV recipients and 5 placebo recipients in each Group. However, due a natural disaster (hurricane Maria), 11 subjects enrolled in Group 1 had loss of samples at key timepoints. To rebalance the number of evaluable subjects between Groups, Group 1 enrollment will be increased by 5 subjects and Group 2 enrollment will be decreased by 5 subjects, for a total enrollment of 50 subjects in Group 1 and 40 in Group 2. Treatment assignments for both groups will be assigned according to the originally planned 8:1 ratio of ZPIV: placebo. Without compromising the blind of the study, we can anticipate approximately 35 evaluable ZPIV recipients and approximately 5 evaluable placebo recipients in each group. All subjects will receive a homologous boost of ZPIV or placebo 28 days post-prime if no halting rules precluding second vaccination are met (Section 9). All subjects will be monitored for occurrence of unsolicited AEs until 28 days after the second vaccination SAEs, AESIs, and history of new medical conditions with onset after the first vaccination will be collected for the duration of the study. Blood for evaluation of antibodies to ZIKV by ELISA and neutralizing antibody assays will be collected at Visit 00, prior to each vaccination, and at multiple timepoints afterward. Primary objectives are: 1) Assess the safety and reactogenicity of a homologous prime boost regimen of ZPIV given at two different dose levels in a dose de-escalation format in healthy adult subjects who live in Puerto Rico, a flavivirus endemic area. 2) Compare the safety and reactogenicity profile of ZPIV after each vaccination, between dosage groups, and by pre-vaccination flavivirus immune status. Secondary Objectives are: 1) Assess the humoral immune response to a homologous prime-boost regimen of ZPIV after each dose of vaccine as determined by kinetics of the immune responses, seroconversion rates, and Geometric Mean Titers (GMT) overall, and compare results between dosage groups and by pre-vaccination flavivirus immune status. 2) Assess the durability of the humoral immune response to ZPIV at 6, 12, 18, and 24 months after the second vaccine administration overall, and compare results between dosage groups and by pre-vaccination flavivirus immune status.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a male or non-pregnant, non-breastfeeding female between the age of 21 and 49 years, inclusive at the time of screening and enrollment.
2. Must be willing and able to read, sign and date the informed consent document before study related procedures are performed.
3. Must be willing and able to comply with study requirements and available for follow-up visits for the entire study.
4. Must have a means to be contacted by telephone.
5. Must have a body mass index (BMI) > /= 18.1 and < 35.0 kg/m2.
6. Must have acceptable* screening laboratory findings within 28 days before enrollment.

   * Acceptable clinical laboratory parameters include:

     * Hemoglobin: women: > /= 11.5 g/dL; men > /= 13.5 g/dL
     * Hemotocrit: women: > /= 34.5%; men > /= 40.5%
     * White blood cell count: > /= 3.500 cells/mm3 but < /= 10,800 cells/mm3
     * Platelets: > /= 150,000 but < /= 450,000 per mm3
     * Urine dipstick (clean urine sample): protein < 1+, glucose negative
     * Serum creatinine < /= 1 x institutional upper limit of normal (ULN)
     * Blood urea nitrogen (BUN) < 25
     * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 1.25 x institutional ULN
     * Total bilirubin < 1.25 x institutional ULN
   * Note: If laboratory screening tests are out of acceptable range, repeat of screening tests is permitted once, provided there is an alternative explanation for the out of range value.
7. Must be in good health based on the investigator's clinical judgment when considering findings from past medical history, medication use, vital signs, and an abbreviated physical examination.

   Note 1: Good health is defined by the absence of any medical condition described in the exclusion criteria in a subject with a normal abbreviated physical exam and vital signs. If the subject has a preexisting condition not listed in exclusion criteria, it cannot meet any of the following criteria: 1) first diagnosed in last 3 months; 2) worsening in terms of clinical outcome in last 6 months; or 3) involves need for medication that may pose a risk to subject's safety or impede assessment of adverse events or immunogenicity if they participate in study.

   Note 2: An abbreviated physical exam differs from a complete exam in that it does not include a genitourinary and rectal exam.

   Note 3: Vital signs must be normal by protocol toxicity grading scale or determined to be normal-variant by investigator. In the event of an abnormal heart rate or blood pressure due to physiological variation or activity, the subject may rest for 10 minutes in a quiet room, and then blood pressure and/or heart rate may be re-measured. Repeated vital signs may be used to determine eligibility.
8. Women of childbearing potential* must have a negative serum pregnancy test at screening and a negative urine pregnancy test immediately prior to each vaccination.

   Note: All female subjects are considered of childbearing potential unless postmenopausal or surgically sterilized and > /= 3 months have passed since sterilization procedure. Postmenopausal is defined as amenorrhea for > /= 12 months without an alternative medical cause. Permanent female sterilization procedures include tubal ligation, bilateral salpingectomy, hysterectomy, bilateral oophorectomy, or successful Essure placement.
9. Women of childbearing potential must use an acceptable method of contraception* from one month (30 days) prior to the first vaccination until the end of the study.

   *Acceptable methods of contraception include the following:
   * Use highly effective contraceptive methods, defined by < 1% failure rate per year independent of user adherence, including long-acting reversible contraception (LARC): progestin-releasing subdermal implants and intrauterine devices (IUD), OR
   * Use effective contraceptive methods, defined by 5-9% failure rate with typical use and < 1% failure rate with consistent and correct use, including: prescription oral contraceptives, contraceptive injections, combined pill, progestin-only pill, hormone-releasing transdermal patch or vaginal ring, and depot medroxyprogesterone acetate injection (Depo-Provera), OR
   * Male sex partners must have had a vasectomy > /= 3 months prior to first vaccination, OR
   * Practice abstinence defined as refraining from heterosexual intercourse from 30 days before first vaccination until the end of the study.
10. Female subjects must agree to not donate eggs (ova, oocytes) from the start of screening period until the end of the study.
11. Subjects must provide concurrent consent at the time of enrollment and 1st vaccination to future use of stored blood samples to measure immunity to ZIKV.

Exclusion Criteria:

1. Has plans to become pregnant during the course of the study, or is currently pregnant or breastfeeding.
2. Plans to receive a licensed flavivirus vaccine or participate in another flavivirus vaccine trial during the study.
3. Has positive serology for HIV 1/2, Hepatitis C virus, or Hepatitis B surface antigen.
4. Has known or suspected congenital or acquired immunodeficiency, or recent history or current use of immunosuppressive therapy* *Anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term (at least 2 weeks within the previous 3 months) systemic corticosteroids therapy (at a dose of at least 0.5 mg/kg/day). Intranasal or topical prednisone (or equivalent) is allowed.
5. Had organ and/or stem cell transplantation whether or not on chronic immunosuppressive therapy.
6. Has history of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure*.

   *Subjects with a history of skin cancer must not be vaccinated at the previous tumor site.
7. Has history of chronic or acute severe neurologic condition*.

   *Including history of Guillain-Barre syndrome, seizure disorder or epilepsy, Bell's palsy, meningitis, or disease with any focal neurologic deficits.
8. Has diabetes mellitus type 1 or type 2, including cases controlled with diet alone.

   *Note: history of isolated gestational diabetes is not an exclusion criterion.
9. Has history of thyroidectomy, or thyroid disease requiring medication during the last 12 months.
10. Has major psychiatric illness during last 12 months that in the investigator's opinion would preclude participation.
11. Has history of other chronic disease or condition*.

    *Includes the conditions and diagnoses defined as AESI in section 9, as well as autoimmune disease, hypercholesterolemia, chronic hepatitis or cirrhosis, chronic pulmonary disease, chronic renal disease, and chronic cardiac disease including hypertension even if medically controlled

    - Vital signs must be normal by protocol toxicity grading scale or determined to be normal-variant by investigator. In the event of an abnormal heart rate or blood pressure due to physiological variation or activity, the subject may rest for 10 minutes in a quiet room, and then blood pressure and/or heart rate may be re-measured. Repeated vital signs may be used to determine eligibility.
12. Has current or past history of substance abuse that in the investigator's opinion would preclude participation.
13. Has tattoos, scars, or other marks on both deltoid areas that would, in the opinion of the investigator, interfere with assessment of the vaccination site.
14. Has a history of chronic urticaria (recurrent hives).
15. Has known allergy or history of anaphylaxis or other serious reaction to a vaccine or vaccine component*.

    *Including aluminum hydroxide (alum) or aminoglycosides (e.g., neomycin and streptomycin).
16. Had major surgery (per the investigator's judgment) in the month prior to screening or plans to have major surgery during the study.
17. Received blood products or immunoglobulin in the 3 months prior to screening or planned use during the course of the study.
18. Donated a unit of blood within 8 weeks before Day 1 or plans to donate blood during the course of the study.
19. Received live attenuated vaccine from 30 days before Day 1 or plans to receive a live attenuated vaccine from Day 1 until 30 days after the last vaccination.
20. Received killed or inactivated vaccine from 14 days before Day 1 or plans to receive a killed or inactivated vaccine from Day 1 until 14 days after the last vaccination.
21. Received experimental therapeutic agents within 3 months prior to the first study vaccination or plans to receive any experimental therapeutic agents during the course of the study.
22. Is currently participating or plans to participate in another clinical study involving an investigational product, blood drawing, or an invasive procedure listed below.

    *An invasive procedure requiring administration of anesthetics or intravenous dyes or removal of tissue would be excluded. This includes endoscopy, bronchoscopy, or administration of IV contrast.
23. Has an acute illness or temperature > /= 38.0ºC on Day 1 or Day 29* or within 2 days prior to vaccination.

    *Subjects with fever or an acute illness on the day of vaccination or in the 2 days prior to vaccination may be re-assessed and enrolled if healthy or only minor residual symptoms remain within 2 days of Day 1 or Day 29.
24. Is a study site employee* or staff paid entirely or partially by the OCRR contract or subcontract for the trial, or staff who are supervised by the PI or Sub-Investigators.

    *Including the Principal Investigator, sub-Investigators listed in Form FDA 1572 or Investigator of Record Form
25. In the investigator's opinion, the subject cannot communicate reliably, is unlikely to adhere to the study requirements, or has a condition that would limit their ability to complete the study.

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ponce School of Medicine CAIMED Center, Ponce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and non-pregnant females between 21 and 49 years old, inclusively. They were recruited from the community at large around the clinic site. The enrollment period occurred between 21MAR2017 and 18JUL2019.
Groups:
- 2.5 mcg ZPIV: 2.5 mcg ZPIV administered intramuscularly in a homologous prime-boost regimen on Day 1 and Day 29. Zika Virus Purified Inactivated Vaccine (ZPIV): Zika Virus Purified Inactivated Vaccine with aluminum hydroxide adjuvant using a 2015 Puerto Rico isolate (PRVABC59 strain).
- 5 mcg ZPIV: 5 mcg ZPIV administered intramuscularly in a homologous prime-boost regimen on Day 1 and Day 29. Zika Virus Purified Inactivated Vaccine (ZPIV): Zika Virus Purified Inactivated Vaccine with aluminum hydroxide adjuvant using a 2015 Puerto Rico isolate (PRVABC59 strain).
- Placebo: Placebo administered intramuscularly on Day 1 and Day 29. Normal saline (0.9% sodium chloride injection, USP) is a clear to colorless, sterile, nonpyrogenic, isotonic solution.
Period: Overall Study
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Started | 36 | 45 | 10
Completed | 26 | 32 | 6
Not Completed | 10 | 13 | 4
Not completed — Physician Decision | 3 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0
Not completed — Lost to Follow-up | 4 | 8 | 3
Not completed — Failure to Meet Randomization Criteria | 1 | 0 | 0
Not completed — Subject Unable to Attend Clinical Visit | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo | Total
Number analyzed (Participants) | 36 | 45 | 10 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (9.0) | 30.5 (8.0) | 28.6 (8.0) | 30.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 25 | 6 | 49
  Male | 18 | 20 | 4 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 45 | 10 | 91
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 15 | 2 | 19
  More than one race | 34 | 18 | 5 | 57
  Unknown or Not Reported | 0 | 12 | 3 | 15
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 36 | 45 | 10 | 91
Baseline ZIKV Immune Status [Count of Participants; unit: Participants]
  Baseline ZIKV Seropositive | 1 | 1 | 0 | 2
  Baseline ZIKV Seronegative | 34 | 43 | 10 | 87
  Unknown | 1 | 1 | 0 | 2
Baseline Flavivirus Immune Status [Count of Participants; unit: Participants]
  Baseline ZIKV Seropositive and DENV Seropositive | 1 | 1 | 0 | 2
  Baseline ZIKV Seropositive and DENV Seronegative | 0 | 0 | 0 | 0
  Baseline ZIKV Seronegative and DENV Seropositive | 26 | 33 | 9 | 68
  Baseline ZIKV Seronegative and DENV Seronegative | 8 | 10 | 1 | 19
  Unknown | 1 | 1 | 0 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.59 (4.09) | 26.51 (3.73) | 29.20 (4.53) | 27.23 (4.01)

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 1 by Treatment Group for All Participants
Description: The following injection site reactogenicity events were measured: pain, tenderness, pruritus, ecchymosis, erythema, and induration. Participants who reported not having a symptom are listed as "None", while participants who did not complete their Memory Aid or could not remember whether they had a symptom are listed as "Not Reported". Severity is the maximum severity reported over all solicited symptoms post dosing for each participant.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- 2.5 mcg ZPIV: 2.5 mcg ZPIV administered intramuscularly in a homologous prime-boost regimen on Day 1 and Day 29.
- 5 mcg ZPIV: 5 mcg ZPIV administered intramuscularly in a homologous prime-boost regimen on Day 1 and Day 29.
- Placebo: Placebo administered intramuscularly on Day 1 and Day 29.
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 35 | 45 | 10
Participants
  Any Local Symptom: None | 15 | 22 | 10
  Any Local Symptom: Mild | 18 | 22 | 0
  Any Local Symptom: Moderate | 2 | 1 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not Reported | 0 | 0 | 0
  Pain: None | 22 | 28 | 10
  Pain: Mild | 11 | 16 | 0
  Pain: Moderate | 2 | 1 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not Reported | 0 | 0 | 0
  Erythema: None | 32 | 45 | 10
  Erythema: Mild | 3 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not Reported | 0 | 0 | 0
  Induration: None | 33 | 44 | 10
  Induration: Mild | 2 | 1 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not Reported | 0 | 0 | 0
  Pruritus: None | 34 | 43 | 10
  Pruritus: Mild | 1 | 2 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not Reported | 0 | 0 | 0
  Ecchymosis: None | 35 | 45 | 10
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not Reported | 0 | 0 | 0
  Tenderness: None | 21 | 29 | 10
  Tenderness: Mild | 13 | 15 | 0
  Tenderness: Moderate | 1 | 1 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not Reported | 0 | 0 | 0

2. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 2 by Treatment Group for All Participants
Description: as for outcome 1
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all participants with available results who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 32 | 43 | 9
Participants
  Any Local Symptom: None | 17 | 33 | 9
  Any Local Symptom: Mild | 15 | 7 | 0
  Any Local Symptom: Moderate | 0 | 3 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not Reported | 0 | 0 | 0
  Pain: None | 20 | 36 | 9
  Pain: Mild | 12 | 4 | 0
  Pain: Moderate | 0 | 3 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not Reported | 0 | 0 | 0
  Erythema: None | 31 | 43 | 9
  Erythema: Mild | 1 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not Reported | 0 | 0 | 0
  Induration: None | 31 | 43 | 9
  Induration: Mild | 1 | 0 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not Reported | 0 | 0 | 0
  Pruritus: None | 30 | 42 | 9
  Pruritus: Mild | 2 | 1 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not Reported | 0 | 0 | 0
  Ecchymosis: None | 32 | 43 | 9
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not Reported | 0 | 0 | 0
  Tenderness: None | 25 | 34 | 9
  Tenderness: Mild | 7 | 6 | 0
  Tenderness: Moderate | 0 | 3 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not Reported | 0 | 0 | 0

3. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 1 by Treatment Group for Baseline ZIKV Seropositive Participants
Description: as for outcome 1
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seropositive participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Any Local Symptom: None | 0 | 1 | 0
  Any Local Symptom: Mild | 1 | 0 | 0
  Any Local Symptom: Moderate | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not reported | 0 | 0 | 0
  Pain: None | 0 | 1 | 0
  Pain: Mild | 1 | 0 | 0
  Pain: Moderate | 0 | 0 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not reported | 0 | 0 | 0
  Erythema: None | 1 | 1 | 0
  Erythema: Mild | 0 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not reported | 0 | 0 | 0
  Induration: None | 1 | 1 | 0
  Induration: Mild | 0 | 0 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not reported | 0 | 0 | 0
  Pruritus: None | 1 | 1 | 0
  Pruritus: Mild | 0 | 0 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not reported | 0 | 0 | 0
  Ecchymosis: None | 1 | 1 | 0
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not reported | 0 | 0 | 0
  Tenderness: None | 1 | 1 | 0
  Tenderness: Mild | 0 | 0 | 0
  Tenderness: Moderate | 0 | 0 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not reported | 0 | 0 | 0

4. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 2 by Treatment Group for Baseline ZIKV Seropositive Participants
Description: as for outcome 1
Time Frame: Day 29 through Day 36
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Any Local Symptom: None | 0 | 1 | 0
  Any Local Symptom: Mild | 1 | 0 | 0
  Any Local Symptom: Moderate | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not reported | 0 | 0 | 0
  Pain: None | 0 | 1 | 0
  Pain: Mild | 1 | 0 | 0
  Pain: Moderate | 0 | 0 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not reported | 0 | 0 | 0
  Erythema: None | 1 | 1 | 0
  Erythema: Mild | 0 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not reported | 0 | 0 | 0
  Induration: None | 1 | 1 | 0
  Induration: Mild | 0 | 0 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not reported | 0 | 0 | 0
  Pruritus: None | 1 | 1 | 0
  Pruritus: Mild | 0 | 0 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not reported | 0 | 0 | 0
  Ecchymosis: None | 1 | 1 | 0
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not reported | 0 | 0 | 0
  Tenderness: None | 0 | 1 | 0
  Tenderness: Mild | 1 | 0 | 0
  Tenderness: Moderate | 0 | 0 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not reported | 0 | 0 | 0

5. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 1 by Treatment Group for Baseline ZIKV Seronegative Participants
Description: as for outcome 1
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seronegative participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 34 | 43 | 10
Participants
  Any Local Symptom: None | 15 | 21 | 10
  Any Local Symptom: Mild | 17 | 21 | 0
  Any Local Symptom: Moderate | 2 | 1 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not Reported | 0 | 0 | 0
  Pain: None | 22 | 27 | 10
  Pain: Mild | 10 | 15 | 0
  Pain: Moderate | 2 | 1 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not Reported | 0 | 0 | 0
  Erythema: None | 31 | 43 | 10
  Erythema: Mild | 3 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not Reported | 0 | 0 | 0
  Induration: None | 32 | 42 | 10
  Induration: Mild | 2 | 1 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not Reported | 0 | 0 | 0
  Pruritus: None | 33 | 41 | 10
  Pruritus: Mild | 1 | 2 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not Reported | 0 | 0 | 0
  Ecchymosis: None | 34 | 43 | 10
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not Reported | 0 | 0 | 0
  Tenderness: None | 20 | 28 | 10
  Tenderness: Mild | 13 | 14 | 0
  Tenderness: Moderate | 1 | 1 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not Reported | 0 | 0 | 0

6. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 2 by Treatment Group for Baseline ZIKV Seronegative Participants
Description: as for outcome 1
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all baseline ZIKV seronegative participants with available results who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 31 | 41 | 9
Participants
  Any Local Symptom: None | 17 | 32 | 9
  Any Local Symptom: Mild | 14 | 6 | 0
  Any Local Symptom: Moderate | 0 | 3 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not Reported | 0 | 0 | 0
  Pain: None | 20 | 34 | 9
  Pain: Mild | 11 | 4 | 0
  Pain: Moderate | 0 | 3 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not Reported | 0 | 0 | 0
  Erythema: None | 30 | 41 | 9
  Erythema: Mild | 1 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not Reported | 0 | 0 | 0
  Induration: None | 30 | 41 | 9
  Induration: Mild | 1 | 0 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not Reported | 0 | 0 | 0
  Pruritus: None | 29 | 40 | 9
  Pruritus: Mild | 2 | 1 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not Reported | 0 | 0 | 0
  Ecchymosis: None | 31 | 41 | 9
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not Reported | 0 | 0 | 0
  Tenderness: None | 25 | 33 | 9
  Tenderness: Mild | 6 | 5 | 0
  Tenderness: Moderate | 0 | 3 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not Reported | 0 | 0 | 0

7. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 1 by Treatment Group for Baseline ZIKV Seropositive and DENV Seropositive Participants
Description: as for outcome 1
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seropositive and DENV seropositive participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Any Local Symptom: None | 0 | 1 | 0
  Any Local Symptom: Mild | 1 | 0 | 0
  Any Local Symptom: Moderate | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not Reported | 0 | 0 | 0
  Pain: None | 0 | 1 | 0
  Pain: Mild | 1 | 0 | 0
  Pain: Moderate | 0 | 0 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not Reported | 0 | 0 | 0
  Erythema: None | 1 | 1 | 0
  Erythema: Mild | 0 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not Reported | 0 | 0 | 0
  Induration: None | 1 | 1 | 0
  Induration: Mild | 0 | 0 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not Reported | 0 | 0 | 0
  Pruritus: None | 1 | 1 | 0
  Pruritus: Mild | 0 | 0 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not Reported | 0 | 0 | 0
  Ecchymosis: None | 1 | 1 | 0
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not Reported | 0 | 0 | 0
  Tenderness: None | 1 | 1 | 0
  Tenderness: Mild | 0 | 0 | 0
  Tenderness: Moderate | 0 | 0 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not Reported | 0 | 0 | 0

8. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 2 by Treatment Group for Baseline ZIKV Seropositive and DENV Seropositive Participants
Description: as for outcome 1
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all baseline ZIKV seropositive and DENV seropositive participants with available results who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Any Local Symptom: None | 0 | 1 | 0
  Any Local Symptom: Mild | 1 | 0 | 0
  Any Local Symptom: Moderate | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not Reported | 0 | 0 | 0
  Pain: None | 0 | 1 | 0
  Pain: Mild | 1 | 0 | 0
  Pain: Moderate | 0 | 0 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not Reported | 0 | 0 | 0
  Erythema: None | 1 | 1 | 0
  Erythema: Mild | 0 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not Reported | 0 | 0 | 0
  Induration: None | 1 | 1 | 0
  Induration: Mild | 0 | 0 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not Reported | 0 | 0 | 0
  Pruritus: None | 1 | 1 | 0
  Pruritus: Mild | 0 | 0 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not Reported | 0 | 0 | 0
  Ecchymosis: None | 1 | 1 | 0
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not Reported | 0 | 0 | 0
  Tenderness: None | 0 | 1 | 0
  Tenderness: Mild | 1 | 0 | 0
  Tenderness: Moderate | 0 | 0 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not Reported | 0 | 0 | 0

9. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 1 by Treatment Group for Baseline ZIKV Seropositive and DENV Seronegative Participants
Description: as for outcome 1
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received at least one study vaccination. No participants met the baseline ZIKV seropositive and DENV seronegative criteria.
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

10. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 2 by Treatment Group for Baseline ZIKV Seropositive and DENV Seronegative Participants
Description: as for outcome 1
Time Frame: Day 29 though Day 36
Population: as for outcome 9
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

11. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 1 by Treatment Group for Baseline ZIKV Seronegative and DENV Seropositive Participants
Description: as for outcome 1
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seronegative and DENV seropositive participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 26 | 33 | 9
Participants
  Any Local Symptom: None | 10 | 17 | 9
  Any Local Symptom: Mild | 14 | 15 | 0
  Any Local Symptom: Moderate | 2 | 1 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not Reported | 0 | 0 | 0
  Pain: None | 17 | 22 | 9
  Pain: Mild | 7 | 10 | 0
  Pain: Moderate | 2 | 1 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not Reported | 0 | 0 | 0
  Erythema: None | 23 | 33 | 9
  Erythema: Mild | 3 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not Reported | 0 | 0 | 0
  Induration: None | 24 | 32 | 9
  Induration: Mild | 2 | 1 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not Reported | 0 | 0 | 0
  Pruritus: None | 25 | 31 | 9
  Pruritus: Mild | 1 | 2 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not Reported | 0 | 0 | 0
  Ecchymosis: None | 26 | 33 | 9
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not Reported | 0 | 0 | 0
  Tenderness: None | 14 | 22 | 9
  Tenderness: Mild | 11 | 10 | 0
  Tenderness: Moderate | 1 | 1 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not Reported | 0 | 0 | 0

12. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 2 by Treatment Group for Baseline ZIKV Seronegative and DENV Seropositive Participants
Description: as for outcome 1
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all baseline ZIKV seronegative and DENV seropositive participants with available results who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 23 | 31 | 8
Participants
  Any Local Symptom: None | 13 | 25 | 8
  Any Local Symptom: Mild | 10 | 3 | 0
  Any Local Symptom: Moderate | 0 | 3 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not Reported | 0 | 0 | 0
  Pain: None | 16 | 26 | 8
  Pain: Mild | 7 | 2 | 0
  Pain: Moderate | 0 | 3 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not Reported | 0 | 0 | 0
  Erythema: None | 22 | 31 | 8
  Erythema: Mild | 1 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not Reported | 0 | 0 | 0
  Induration: None | 22 | 31 | 8
  Induration: Mild | 1 | 0 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not Reported | 0 | 0 | 0
  Pruritus: None | 22 | 30 | 8
  Pruritus: Mild | 1 | 1 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not Reported | 0 | 0 | 0
  Ecchymosis: None | 23 | 31 | 8
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not Reported | 0 | 0 | 0
  Tenderness: None | 18 | 26 | 8
  Tenderness: Mild | 5 | 2 | 0
  Tenderness: Moderate | 0 | 3 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not Reported | 0 | 0 | 0

13. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 1 by Treatment Group for Baseline ZIKV Seronegative and DENV Seronegative Participants
Description: as for outcome 1
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seronegative and DENV seronegative participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 8 | 10 | 1
Participants
  Any Local Symptom: None | 5 | 4 | 1
  Any Local Symptom: Mild | 3 | 6 | 0
  Any Local Symptom: Moderate | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not Reported | 0 | 0 | 0
  Pain: None | 5 | 5 | 1
  Pain: Mild | 3 | 5 | 0
  Pain: Moderate | 0 | 0 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not Reported | 0 | 0 | 0
  Erythema: None | 8 | 10 | 1
  Erythema: Mild | 0 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not Reported | 0 | 0 | 0
  Induration: None | 8 | 10 | 1
  Induration: Mild | 0 | 0 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not Reported | 0 | 0 | 0
  Pruritus: None | 8 | 10 | 1
  Pruritus: Mild | 0 | 0 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not Reported | 0 | 0 | 0
  Ecchymosis: None | 8 | 10 | 1
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not Reported | 0 | 0 | 0
  Tenderness: None | 6 | 6 | 1
  Tenderness: Mild | 2 | 4 | 0
  Tenderness: Moderate | 0 | 0 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not Reported | 0 | 0 | 0

14. Primary Outcome: Frequency and Severity of Solicited Local Events Post Dose 2 by Treatment Group for Baseline ZIKV Seronegative and DENV Seronegative Participants
Description: as for outcome 1
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all baseline ZIKV seronegative and DENV seronegative participants with available results who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 8 | 10 | 1
Participants
  Any Local Symptom: None | 4 | 7 | 1
  Any Local Symptom: Mild | 4 | 3 | 0
  Any Local Symptom: Moderate | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0
  Any Local Symptom: Not Reported | 0 | 0 | 0
  Pain: None | 4 | 8 | 1
  Pain: Mild | 4 | 2 | 0
  Pain: Moderate | 0 | 0 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Not Reported | 0 | 0 | 0
  Erythema: None | 8 | 10 | 1
  Erythema: Mild | 0 | 0 | 0
  Erythema: Moderate | 0 | 0 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Not Reported | 0 | 0 | 0
  Induration: None | 8 | 10 | 1
  Induration: Mild | 0 | 0 | 0
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Induration: Not Reported | 0 | 0 | 0
  Pruritus: None | 7 | 10 | 1
  Pruritus: Mild | 1 | 0 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: Not Reported | 0 | 0 | 0
  Ecchymosis: None | 8 | 10 | 1
  Ecchymosis: Mild | 0 | 0 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Ecchymosis: Not Reported | 0 | 0 | 0
  Tenderness: None | 7 | 7 | 1
  Tenderness: Mild | 1 | 3 | 0
  Tenderness: Moderate | 0 | 0 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Not Reported | 0 | 0 | 0

15. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 1 by Treatment Group for All Participants
Description: The following systemic solicited events were measured: feverishness, fatigue, malaise, myalgia, arthralgia, headache, nausea, vomiting, diarrhea, abdominal pain, rash, and fever. Participants who reported not having a symptom are listed as "None", while participants who did not complete their Memory Aid or could not remember whether they had a symptom are listed as "Not Reported". Severity is the maximum severity reported over all solicited symptoms post dosing for each participant.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 35 | 45 | 10
Participants
  Any Systemic Symptom: None | 21 | 25 | 5
  Any Systemic Symptom: Mild | 11 | 17 | 4
  Any Systemic Symptom: Moderate | 3 | 3 | 1
  Any Systemic Symptom: Severe | 0 | 0 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 33 | 43 | 9
  Feverishness: Mild | 2 | 2 | 0
  Feverishness: Moderate | 0 | 0 | 1
  Feverishness: Severe | 0 | 0 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 32 | 37 | 6
  Fatigue: Mild | 2 | 7 | 3
  Fatigue: Moderate | 1 | 1 | 1
  Fatigue: Severe | 0 | 0 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 32 | 43 | 9
  Malaise: Mild | 3 | 2 | 1
  Malaise: Moderate | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Myalgia: None | 30 | 41 | 8
  Myalgia: Mild | 4 | 3 | 1
  Myalgia: Moderate | 1 | 1 | 1
  Myalgia: Severe | 0 | 0 | 0
  Myalgia: Not Reported | 0 | 0 | 0
  Arthralgia: None | 32 | 42 | 9
  Arthralgia: Mild | 3 | 3 | 0
  Arthralgia: Moderate | 0 | 0 | 1
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 25 | 33 | 6
  Headache: Mild | 9 | 11 | 3
  Headache: Moderate | 1 | 1 | 1
  Headache: Severe | 0 | 0 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 33 | 40 | 10
  Nausea: Mild | 2 | 5 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 34 | 45 | 10
  Vomiting: Mild | 1 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 35 | 43 | 10
  Diarrhea: Mild | 0 | 2 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 35 | 44 | 10
  Abdominal Pain: Mild | 0 | 1 | 0
  Abdominal Pain: Moderate | 0 | 0 | 0
  Abdominal Pain: Severe | 0 | 0 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 34 | 45 | 10
  Rash: Mild | 1 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 34 | 44 | 9
  Fever: Mild | 1 | 1 | 0
  Fever: Moderate | 0 | 0 | 1
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

16. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 2 by Treatment Group for All Participants
Description: as for outcome 15
Time Frame: Day 29 through Day 36
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 32 | 43 | 9
Participants
  Any Systemic Symptom: None | 26 | 36 | 8
  Any Systemic Symptom: Mild | 5 | 5 | 1
  Any Systemic Symptom: Moderate | 1 | 1 | 0
  Any Systemic Symptom: Severe | 0 | 1 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 32 | 42 | 9
  Feverishness: Mild | 0 | 0 | 0
  Feverishness: Moderate | 0 | 0 | 0
  Feverishness: Severe | 0 | 1 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 31 | 40 | 9
  Fatigue: Mild | 1 | 1 | 0
  Fatigue: Moderate | 0 | 1 | 0
  Fatigue: Severe | 0 | 1 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 31 | 40 | 9
  Malaise: Mild | 1 | 1 | 0
  Malaise: Moderate | 0 | 1 | 0
  Malaise: Severe | 0 | 1 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Myalgia: None | 30 | 39 | 9
  Myalgia: Mild | 2 | 2 | 0
  Myalgia: Moderate | 0 | 1 | 0
  Myalgia: Severe | 0 | 1 | 0
  Myalgia: Not Reported | 0 | 0 | 0
  Arthralgia: None | 32 | 41 | 9
  Arthralgia: Mild | 0 | 0 | 0
  Arthralgia: Moderate | 0 | 1 | 0
  Arthralgia: Severe | 0 | 1 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 26 | 39 | 8
  Headache: Mild | 6 | 3 | 1
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 1 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 30 | 41 | 9
  Nausea: Mild | 2 | 1 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 1 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 32 | 42 | 9
  Vomiting: Mild | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 1 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 32 | 42 | 9
  Diarrhea: Mild | 0 | 1 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 31 | 42 | 9
  Abdominal Pain: Mild | 0 | 0 | 0
  Abdominal Pain: Moderate | 1 | 0 | 0
  Abdominal Pain: Severe | 0 | 1 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 32 | 43 | 9
  Rash: Mild | 0 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 32 | 41 | 9
  Fever: Mild | 0 | 1 | 0
  Fever: Moderate | 0 | 1 | 0
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

17. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 1 by Treatment Group for Baseline ZIKV Seropositive Participants
Description: as for outcome 15
Time Frame: Day 1 through Day 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Any Systemic Symptom: None | 0 | 1 | 0
  Any Systemic Symptom: Mild | 1 | 0 | 0
  Any Systemic Symptom: Moderate | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 1 | 1 | 0
  Feverishness: Mild | 0 | 0 | 0
  Feverishness: Moderate | 0 | 0 | 0
  Feverishness: Severe | 0 | 0 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 0 | 1 | 0
  Fatigue: Mild | 1 | 0 | 0
  Fatigue: Moderate | 0 | 0 | 0
  Fatigue: Severe | 0 | 0 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 1 | 1 | 0
  Malaise: Mild | 0 | 0 | 0
  Malaise: Moderate | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Arthralgia: None | 1 | 1 | 0
  Arthralgia: Mild | 0 | 0 | 0
  Arthralgia: Moderate | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 1 | 1 | 0
  Headache: Mild | 0 | 0 | 0
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 1 | 1 | 0
  Nausea: Mild | 0 | 0 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 1 | 1 | 0
  Vomiting: Mild | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 1 | 1 | 0
  Diarrhea: Mild | 0 | 0 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 1 | 1 | 0
  Abdominal Pain: Mild | 0 | 0 | 0
  Abdominal Pain: Moderate | 0 | 0 | 0
  Abdominal Pain: Severe | 0 | 0 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 1 | 1 | 0
  Rash: Mild | 0 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 1 | 1 | 0
  Fever: Mild | 0 | 0 | 0
  Fever: Moderate | 0 | 0 | 0
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

18. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 2 by Treatment Group for Baseline ZIKV Seropositive Participants
Description: as for outcome 15
Time Frame: Day 29 through Day 36
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Any Systemic Symptom: None | 1 | 1 | 0
  Any Systemic Symptom: Mild | 0 | 0 | 0
  Any Systemic Symptom: Moderate | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 1 | 1 | 0
  Feverishness: Mild | 0 | 0 | 0
  Feverishness: Moderate | 0 | 0 | 0
  Feverishness: Severe | 0 | 0 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 1 | 1 | 0
  Fatigue: Mild | 0 | 0 | 0
  Fatigue: Moderate | 0 | 0 | 0
  Fatigue: Severe | 0 | 0 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 1 | 1 | 0
  Malaise: Mild | 0 | 0 | 0
  Malaise: Moderate | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Myalgia: None | 1 | 1 | 0
  Myalgia: Mild | 0 | 0 | 0
  Myalgia: Moderate | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0
  Myalgia: Not Reported | 0 | 0 | 0
  Arthralgia: None | 1 | 1 | 0
  Arthralgia: Mild | 0 | 0 | 0
  Arthralgia: Moderate | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 1 | 1 | 0
  Headache: Mild | 0 | 0 | 0
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 1 | 1 | 0
  Nausea: Mild | 0 | 0 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 1 | 1 | 0
  Vomiting: Mild | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 1 | 1 | 0
  Diarrhea: Mild | 0 | 0 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 1 | 1 | 0
  Abdominal Pain: Mild | 0 | 0 | 0
  Abdominal Pain: Moderate | 0 | 0 | 0
  Abdominal Pain: Severe | 0 | 0 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 1 | 1 | 0
  Rash: Mild | 0 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 1 | 1 | 0
  Fever: Mild | 0 | 0 | 0
  Fever: Moderate | 0 | 0 | 0
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

19. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 1 by Treatment Group for Baseline ZIKV Seronegative Participants
Description: as for outcome 15
Time Frame: Day 1 through Day 8
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 34 | 43 | 10
Participants
  Any Systemic Symptom: None | 21 | 24 | 5
  Any Systemic Symptom: Mild | 10 | 17 | 4
  Any Systemic Symptom: Moderate | 3 | 2 | 1
  Any Systemic Symptom: Severe | 0 | 0 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 32 | 42 | 9
  Feverishness: Mild | 2 | 1 | 0
  Feverishness: Moderate | 0 | 0 | 1
  Feverishness: Severe | 0 | 0 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 32 | 36 | 6
  Fatigue: Mild | 1 | 6 | 3
  Fatigue: Moderate | 1 | 1 | 1
  Fatigue: Severe | 0 | 0 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 31 | 42 | 9
  Malaise: Mild | 3 | 1 | 1
  Malaise: Moderate | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Myalgia: None | 29 | 40 | 8
  Myalgia: Mild | 4 | 3 | 1
  Myalgia: Moderate | 1 | 0 | 1
  Myalgia: Severe | 0 | 0 | 0
  Myalgia: Not Reported | 0 | 0 | 0
  Arthralgia: None | 31 | 41 | 9
  Arthralgia: Mild | 3 | 2 | 0
  Arthralgia: Moderate | 0 | 0 | 1
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 24 | 32 | 6
  Headache: Mild | 9 | 10 | 3
  Headache: Moderate | 1 | 1 | 1
  Headache: Severe | 0 | 0 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 32 | 38 | 10
  Nausea: Mild | 2 | 5 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 33 | 43 | 10
  Vomiting: Mild | 1 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 34 | 41 | 10
  Diarrhea: Mild | 0 | 2 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 34 | 43 | 10
  Abdominal Pain: Mild | 0 | 0 | 0
  Abdominal Pain: Moderate | 0 | 0 | 0
  Abdominal Pain: Severe | 0 | 0 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 33 | 43 | 10
  Rash: Mild | 1 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 33 | 42 | 9
  Fever: Mild | 1 | 1 | 0
  Fever: Moderate | 0 | 0 | 1
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

20. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 2 by Treatment Group for Baseline ZIKV Seronegative Participants
Description: as for outcome 15
Time Frame: Day 29 through Day 36
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 31 | 41 | 9
Participants
  Any Systemic Symptom: None | 25 | 35 | 8
  Any Systemic Symptom: Mild | 5 | 4 | 1
  Any Systemic Symptom: Moderate | 1 | 1 | 0
  Any Systemic Symptom: Severe | 0 | 1 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 31 | 40 | 9
  Feverishness: Mild | 0 | 0 | 0
  Feverishness: Moderate | 0 | 0 | 0
  Feverishness: Severe | 0 | 1 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 30 | 38 | 9
  Fatigue: Mild | 1 | 1 | 0
  Fatigue: Moderate | 0 | 1 | 0
  Fatigue: Severe | 0 | 1 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 30 | 38 | 9
  Malaise: Mild | 1 | 1 | 0
  Malaise: Moderate | 0 | 1 | 0
  Malaise: Severe | 0 | 1 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Myalgia: None | 29 | 38 | 9
  Myalgia: Mild | 2 | 1 | 0
  Myalgia: Moderate | 0 | 1 | 0
  Myalgia: Severe | 0 | 1 | 0
  Myalgia: Not Reported | 0 | 0 | 0
  Arthralgia: None | 31 | 39 | 9
  Arthralgia: Mild | 0 | 0 | 0
  Arthralgia: Moderate | 0 | 1 | 0
  Arthralgia: Severe | 0 | 1 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 25 | 37 | 8
  Headache: Mild | 6 | 3 | 1
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 1 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 29 | 39 | 9
  Nausea: Mild | 2 | 1 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 1 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 31 | 40 | 9
  Vomiting: Mild | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 1 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 31 | 40 | 9
  Diarrhea: Mild | 0 | 1 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 30 | 40 | 9
  Abdominal Pain: Mild | 0 | 0 | 0
  Abdominal Pain: Moderate | 1 | 0 | 0
  Abdominal Pain: Severe | 0 | 1 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 31 | 41 | 9
  Rash: Mild | 0 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 31 | 39 | 9
  Fever: Mild | 0 | 1 | 0
  Fever: Moderate | 0 | 1 | 0
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

21. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 1 by Treatment Group for Baseline ZIKV Seropositive and DENV Seropositive Participants
Description: as for outcome 15
Time Frame: Day 1 through Day 8
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Any Systemic Symptom: None | 0 | 1 | 0
  Any Systemic Symptom: Mild | 1 | 0 | 0
  Any Systemic Symptom: Moderate | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 1 | 1 | 0
  Feverishness: Mild | 0 | 0 | 0
  Feverishness: Moderate | 0 | 0 | 0
  Feverishness: Severe | 0 | 0 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 0 | 1 | 0
  Fatigue: Mild | 1 | 0 | 0
  Fatigue: Moderate | 0 | 0 | 0
  Fatigue: Severe | 0 | 0 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 1 | 1 | 0
  Malaise: Mild | 0 | 0 | 0
  Malaise: Moderate | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Myalgia: None | 1 | 1 | 0
  Myalgia: Mild | 0 | 0 | 0
  Myalgia: Moderate | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0
  Myalgia: Not Reported | 0 | 0 | 0
  Arthralgia: None | 1 | 1 | 0
  Arthralgia: Mild | 0 | 0 | 0
  Arthralgia: Moderate | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 1 | 1 | 0
  Headache: Mild | 0 | 0 | 0
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 1 | 1 | 0
  Nausea: Mild | 0 | 0 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 1 | 1 | 0
  Vomiting: Mild | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 1 | 1 | 0
  Diarrhea: Mild | 0 | 0 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 1 | 1 | 0
  Abdominal Pain: Mild | 0 | 0 | 0
  Abdominal Pain: Moderate | 0 | 0 | 0
  Abdominal Pain: Severe | 0 | 0 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 1 | 1 | 0
  Rash: Mild | 0 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 1 | 1 | 0
  Fever: Mild | 0 | 0 | 0
  Fever: Moderate | 0 | 0 | 0
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

22. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 2 by Treatment Group for Baseline ZIKV Seropositive and DENV Seropositive Participants
Description: as for outcome 15
Time Frame: Day 29 through Day 36
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Any Systemic Symptom: None | 1 | 1 | 0
  Any Systemic Symptom: Mild | 0 | 0 | 0
  Any Systemic Symptom: Moderate | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 1 | 1 | 0
  Feverishness: Mild | 0 | 0 | 0
  Feverishness: Moderate | 0 | 0 | 0
  Feverishness: Severe | 0 | 0 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 1 | 1 | 0
  Fatigue: Mild | 0 | 0 | 0
  Fatigue: Moderate | 0 | 0 | 0
  Fatigue: Severe | 0 | 0 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 1 | 1 | 0
  Malaise: Mild | 0 | 0 | 0
  Malaise: Moderate | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Myalgia: None | 1 | 1 | 0
  Myalgia: Mild | 0 | 0 | 0
  Myalgia: Moderate | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0
  Myalgia: Not Reported | 0 | 0 | 0
  Arthralgia: None | 1 | 1 | 0
  Arthralgia: Mild | 0 | 0 | 0
  Arthralgia: Moderate | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 1 | 1 | 0
  Headache: Mild | 0 | 0 | 0
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 1 | 1 | 0
  Nausea: Mild | 0 | 0 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 1 | 1 | 0
  Vomiting: Mild | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 1 | 1 | 0
  Diarrhea: Mild | 0 | 0 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 1 | 1 | 0
  Abdominal Pain: Mild | 0 | 0 | 0
  Abdominal Pain: Moderate | 0 | 0 | 0
  Abdominal Pain: Severe | 0 | 0 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 1 | 1 | 0
  Rash: Mild | 0 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 1 | 1 | 0
  Fever: Mild | 0 | 0 | 0
  Fever: Moderate | 0 | 0 | 0
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

23. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 1 by Treatment Group for Baseline ZIKV Seropositive and DENV Seronegative Participants
Description: as for outcome 15
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seropositive and DENV seronegative participants who received at least one study vaccination. No subjects met the baseline ZIKV seropositive and DENV seronegative criteria.
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

24. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 2 by Treatment Group for Baseline ZIKV Seropositive and DENV Seronegative Participants
Description: as for outcome 15
Time Frame: Day 29 through Day 36
Population: as for outcome 23
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

25. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 1 by Treatment Group for Baseline ZIKV Seronegative and DENV Seropositive Participants
Description: as for outcome 15
Time Frame: Day 1 through Day 8
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 26 | 33 | 9
Participants
  Any Systemic Symptom: None | 17 | 18 | 5
  Any Systemic Symptom: Mild | 7 | 13 | 3
  Any Systemic Symptom: Moderate | 2 | 2 | 1
  Any Systemic Symptom: Severe | 0 | 0 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 25 | 33 | 8
  Feverishness: Mild | 1 | 0 | 0
  Feverishness: Moderate | 0 | 0 | 1
  Feverishness: Severe | 0 | 0 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 25 | 27 | 5
  Fatigue: Mild | 1 | 5 | 3
  Fatigue: Moderate | 0 | 1 | 1
  Fatigue: Severe | 0 | 0 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 23 | 32 | 8
  Malaise: Mild | 3 | 1 | 1
  Malaise: Moderate | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Myalgia: None | 22 | 30 | 7
  Myalgia: Mild | 3 | 3 | 1
  Myalgia: Moderate | 1 | 0 | 1
  Myalgia: Severe | 0 | 0 | 0
  Myalgia: Not Reported | 0 | 0 | 0
  Arthralgia: None | 23 | 32 | 8
  Arthralgia: Mild | 3 | 1 | 0
  Arthralgia: Moderate | 0 | 0 | 1
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 19 | 23 | 6
  Headache: Mild | 6 | 9 | 2
  Headache: Moderate | 1 | 1 | 1
  Headache: Severe | 0 | 0 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 24 | 29 | 9
  Nausea: Mild | 2 | 4 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 25 | 33 | 9
  Vomiting: Mild | 1 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 26 | 32 | 9
  Diarrhea: Mild | 0 | 1 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 26 | 33 | 9
  Abdominal Pain: Mild | 0 | 0 | 0
  Abdominal Pain: Moderate | 0 | 0 | 0
  Abdominal Pain: Severe | 0 | 0 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 25 | 33 | 9
  Rash: Mild | 1 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 25 | 32 | 8
  Fever: Mild | 1 | 1 | 0
  Fever: Moderate | 0 | 0 | 1
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

26. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 2 by Treatment Group for Baseline ZIKV Seronegative and DENV Seropositive Participants
Description: as for outcome 15
Time Frame: Day 29 through Day 36
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 23 | 31 | 8
Participants
  Any Systemic Symptom: None | 19 | 27 | 8
  Any Systemic Symptom: Mild | 3 | 3 | 0
  Any Systemic Symptom: Moderate | 1 | 1 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 23 | 31 | 8
  Feverishness: Mild | 0 | 0 | 0
  Feverishness: Moderate | 0 | 0 | 0
  Feverishness: Severe | 0 | 0 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 22 | 30 | 8
  Fatigue: Mild | 1 | 0 | 0
  Fatigue: Moderate | 0 | 1 | 0
  Fatigue: Severe | 0 | 0 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 22 | 30 | 8
  Malaise: Mild | 1 | 0 | 0
  Malaise: Moderate | 0 | 1 | 0
  Malaise: Severe | 0 | 0 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Myalgia: None | 22 | 30 | 8
  Myalgia: Mild | 1 | 0 | 0
  Myalgia: Moderate | 0 | 1 | 0
  Myalgia: Severe | 0 | 0 | 0
  Myalgia: Not Reported | 0 | 0 | 0
  Arthralgia: None | 23 | 30 | 8
  Arthralgia: Mild | 0 | 0 | 0
  Arthralgia: Moderate | 0 | 1 | 0
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 19 | 29 | 8
  Headache: Mild | 4 | 2 | 0
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 22 | 30 | 8
  Nausea: Mild | 1 | 1 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 23 | 31 | 8
  Vomiting: Mild | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 23 | 31 | 8
  Diarrhea: Mild | 0 | 0 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 22 | 31 | 8
  Abdominal Pain: Mild | 0 | 0 | 0
  Abdominal Pain: Moderate | 1 | 0 | 0
  Abdominal Pain: Severe | 0 | 0 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 23 | 31 | 8
  Rash: Mild | 0 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 23 | 30 | 8
  Fever: Mild | 0 | 1 | 0
  Fever: Moderate | 0 | 0 | 0
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

27. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 1 by Treatment Group for Baseline ZIKV Seronegative and DENV Seronegative Participants
Description: as for outcome 15
Time Frame: Day 1 through Day 8
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 8 | 10 | 1
Participants
  Any Systemic Symptom: None | 4 | 6 | 0
  Any Systemic Symptom: Mild | 3 | 4 | 1
  Any Systemic Symptom: Moderate | 1 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 7 | 9 | 1
  Feverishness: Mild | 1 | 1 | 0
  Feverishness: Moderate | 0 | 0 | 0
  Feverishness: Severe | 0 | 0 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 7 | 9 | 1
  Fatigue: Mild | 0 | 1 | 0
  Fatigue: Moderate | 1 | 0 | 0
  Fatigue: Severe | 0 | 0 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 8 | 10 | 1
  Malaise: Mild | 0 | 0 | 0
  Malaise: Moderate | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Myalgia: None | 7 | 10 | 1
  Myalgia: Mild | 1 | 0 | 0
  Myalgia: Moderate | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0
  Myalgia: Not Reported | 0 | 0 | 0
  Arthralgia: None | 8 | 9 | 1
  Arthralgia: Mild | 0 | 1 | 0
  Arthralgia: Moderate | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 5 | 9 | 0
  Headache: Mild | 3 | 1 | 1
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 8 | 9 | 1
  Nausea: Mild | 0 | 1 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 8 | 10 | 1
  Vomiting: Mild | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 8 | 9 | 1
  Diarrhea: Mild | 0 | 1 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 8 | 10 | 1
  Abdominal Pain: Mild | 0 | 0 | 0
  Abdominal Pain: Moderate | 0 | 0 | 0
  Abdominal Pain: Severe | 0 | 0 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 8 | 10 | 1
  Rash: Mild | 0 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 8 | 10 | 1
  Fever: Mild | 0 | 0 | 0
  Fever: Moderate | 0 | 0 | 0
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

28. Primary Outcome: Frequency and Severity of Solicited Systemic Events Post Dose 2 by Treatment Group for Baseline ZIKV Seronegative and DENV Seronegative Participants
Description: as for outcome 15
Time Frame: Day 29 through Day 36
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 8 | 10 | 1
Participants
  Any Systemic Symptom: None | 6 | 8 | 0
  Any Systemic Symptom: Mild | 2 | 1 | 1
  Any Systemic Symptom: Moderate | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 1 | 0
  Any Systemic Symptom: Not Reported | 0 | 0 | 0
  Feverishness: None | 8 | 9 | 1
  Feverishness: Mild | 0 | 0 | 0
  Feverishness: Moderate | 0 | 0 | 0
  Feverishness: Severe | 0 | 1 | 0
  Feverishness: Not Reported | 0 | 0 | 0
  Fatigue: None | 8 | 8 | 1
  Fatigue: Mild | 0 | 1 | 0
  Fatigue: Moderate | 0 | 0 | 0
  Fatigue: Severe | 0 | 1 | 0
  Fatigue: Not Reported | 0 | 0 | 0
  Malaise: None | 8 | 8 | 1
  Malaise: Mild | 0 | 1 | 0
  Malaise: Moderate | 0 | 0 | 0
  Malaise: Severe | 0 | 1 | 0
  Malaise: Not Reported | 0 | 0 | 0
  Myalgia: None | 7 | 8 | 1
  Myalgia: Mild | 1 | 1 | 0
  Myalgia: Moderate | 0 | 0 | 0
  Myalgia: Severe | 0 | 1 | 0
  Myalgia: Not Reported | 0 | 0 | 0
  Arthralgia: None | 8 | 9 | 1
  Arthralgia: Mild | 0 | 0 | 0
  Arthralgia: Moderate | 0 | 0 | 0
  Arthralgia: Severe | 0 | 1 | 0
  Arthralgia: Not Reported | 0 | 0 | 0
  Headache: None | 6 | 8 | 0
  Headache: Mild | 2 | 1 | 1
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 1 | 0
  Headache: Not Reported | 0 | 0 | 0
  Nausea: None | 7 | 9 | 1
  Nausea: Mild | 1 | 0 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 1 | 0
  Nausea: Not Reported | 0 | 0 | 0
  Vomiting: None | 8 | 9 | 1
  Vomiting: Mild | 0 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 1 | 0
  Vomiting: Not Reported | 0 | 0 | 0
  Diarrhea: None | 8 | 9 | 1
  Diarrhea: Mild | 0 | 1 | 0
  Diarrhea: Moderate | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0
  Diarrhea: Not Reported | 0 | 0 | 0
  Abdominal Pain: None | 8 | 9 | 1
  Abdominal Pain: Mild | 0 | 0 | 0
  Abdominal Pain: Moderate | 0 | 0 | 0
  Abdominal Pain: Severe | 0 | 1 | 0
  Abdominal Pain: Not Reported | 0 | 0 | 0
  Rash: None | 8 | 10 | 1
  Rash: Mild | 0 | 0 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0
  Rash: Not Reported | 0 | 0 | 0
  Fever: None | 8 | 9 | 1
  Fever: Mild | 0 | 0 | 0
  Fever: Moderate | 0 | 1 | 0
  Fever: Severe | 0 | 0 | 0
  Fever: Not Reported | 0 | 0 | 0

29. Primary Outcome: Frequency and Severity of Unsolicited Adverse Events by Treatment Group for All Participants
Description: Adverse events (AEs) are defined as any untoward medical occurrence regardless of its causal relationship to study treatment. Number of participants with an AE are summarized by MedDRA System Organ Class (SOC). If a condition was present at screening, it was not considered an AE unless the severity worsened.
Time Frame: Day 1 through Day 57
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 35 | 45 | 10
Participants
  Any SOC: Mild | 21 | 27 | 5
  Any SOC: Moderate | 6 | 12 | 0
  Any SOC: Severe | 2 | 4 | 1
  Cardiac Disorders : Mild | 0 | 3 | 0
  Cardiac Disorders : Moderate | 0 | 1 | 0
  Cardiac Disorders : Severe | 0 | 0 | 0
  Eye Disorders : Mild | 1 | 2 | 0
  Eye Disorders : Moderate | 1 | 1 | 0
  Eye Disorders : Severe | 0 | 1 | 0
  Gastrointestinal Disorders : Mild | 4 | 1 | 0
  Gastrointestinal Disorders : Moderate | 0 | 2 | 0
  Gastrointestinal Disorders : Severe | 0 | 1 | 0
  General Disorders and Administration Site Conditions : Mild | 2 | 2 | 1
  General Disorders and Administration Site Conditions : Moderate | 1 | 3 | 0
  General Disorders and Administration Site Conditions : Severe | 1 | 2 | 0
  Immune System Disorders : Mild | 0 | 0 | 0
  Immune System Disorders : Moderate | 0 | 1 | 0
  Immune System Disorders : Severe | 0 | 0 | 0
  Infections and Infestations : Mild | 9 | 9 | 3
  Infections and Infestations : Moderate | 2 | 2 | 0
  Infections and Infestations : Severe | 0 | 4 | 0
  Injury, Poisoning and Procedural Complications : Mild | 1 | 4 | 0
  Injury, Poisoning and Procedural Complications : Moderate | 1 | 1 | 0
  Injury, Poisoning and Procedural Complications : Severe | 0 | 0 | 1
  Investigations : Mild | 4 | 4 | 0
  Investigations : Moderate | 0 | 0 | 0
  Investigations : Severe | 0 | 0 | 0
  Metabolism and nutrition disorders: Mild | 1 | 0 | 0
  Metabolism and nutrition disorders: Moderate | 0 | 0 | 0
  Metabolism and nutrition disorders: Severe | 0 | 0 | 0
  Musculoskeletal and Connective Tissue Disorders : Mild | 2 | 1 | 0
  Musculoskeletal and Connective Tissue Disorders : Moderate | 0 | 4 | 0
  Musculoskeletal and Connective Tissue Disorders : Severe | 1 | 3 | 0
  Nervous System Disorders : Mild | 2 | 3 | 2
  Nervous System Disorders : Moderate | 3 | 3 | 0
  Nervous System Disorders : Severe | 2 | 2 | 0
  Psychiatric disorders: Mild | 2 | 0 | 0
  Psychiatric disorders: Moderate | 1 | 0 | 0
  Psychiatric disorders: Severe | 0 | 0 | 0
  Renal and urinary disorders: Mild | 1 | 0 | 0
  Renal and urinary disorders: Moderate | 0 | 0 | 0
  Renal and urinary disorders: Severe | 0 | 0 | 0
  Reproductive System and Breast Disorders : Mild | 0 | 1 | 0
  Reproductive System and Breast Disorders : Moderate | 0 | 1 | 0
  Reproductive System and Breast Disorders : Severe | 0 | 0 | 0
  Respiratory, Thoracic, and Mediastinal Disorders : Mild | 4 | 1 | 1
  Respiratory, Thoracic, and Mediastinal Disorders : Moderate | 0 | 0 | 0
  Respiratory, Thoracic, and Mediastinal Disorders : Severe | 0 | 0 | 0
  Skin and Subcutaneous Tissue Disorders : Mild | 3 | 7 | 1
  Skin and Subcutaneous Tissue Disorders : Moderate | 0 | 2 | 0
  Skin and Subcutaneous Tissue Disorders : Severe | 1 | 0 | 0

30. Primary Outcome: Frequency and Severity of Unsolicited Adverse Events by Treatment Group for Baseline ZIKV Seropositive Participants
Description: as for outcome 29
Time Frame: Day 1 through Day 57
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Any SOC: Mild | 0 | 0 | 0
  Any SOC: Moderate | 1 | 0 | 0
  Any SOC: Severe | 0 | 0 | 0
  Infections and infestations: Mild | 0 | 0 | 0
  Infections and infestations: Moderate | 1 | 0 | 0
  Infections and infestations: Severe | 0 | 0 | 0

31. Primary Outcome: Frequency and Severity of Unsolicited Adverse Events by Treatment Group for Baseline ZIKV Seronegative Participants
Description: as for outcome 29
Time Frame: Day 1 through Day 57
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 34 | 43 | 10
Participants
  Any SOC : Mild | 21 | 26 | 5
  Any SOC : Moderate | 5 | 11 | 0
  Any SOC : Severe | 2 | 4 | 1
  Cardiac disorders : Mild | 0 | 3 | 0
  Cardiac disorders : Moderate | 0 | 1 | 0
  Cardiac disorders : Severe | 0 | 0 | 0
  Eye disorders : Mild | 1 | 2 | 0
  Eye disorders : Moderate | 1 | 1 | 0
  Eye disorders : Severe | 0 | 1 | 0
  Gastrointestinal disorders : Mild | 4 | 1 | 0
  Gastrointestinal disorders : Moderate | 0 | 1 | 0
  Gastrointestinal disorders : Severe | 0 | 1 | 0
  General disorders and administration site conditions : Mild | 2 | 2 | 1
  General disorders and administration site conditions : Moderate | 1 | 3 | 0
  General disorders and administration site conditions : Severe | 1 | 2 | 0
  Immune system disorders : Mild | 0 | 0 | 0
  Immune system disorders : Moderate | 0 | 1 | 0
  Immune system disorders : Severe | 0 | 0 | 0
  Infections and infestations : Mild | 9 | 8 | 3
  Infections and infestations : Moderate | 1 | 2 | 0
  Infections and infestations : Severe | 0 | 4 | 0
  Injury, poisoning and procedural complications : Mild | 1 | 4 | 0
  Injury, poisoning and procedural complications : Moderate | 1 | 1 | 0
  Injury, poisoning and procedural complications : Severe | 0 | 0 | 1
  Investigations : Mild | 4 | 4 | 0
  Investigations : Moderate | 0 | 0 | 0
  Investigations : Severe | 0 | 0 | 0
  Metabolism and nutrition disorders: Mild | 1 | 0 | 0
  Metabolism and nutrition disorders: Moderate | 0 | 0 | 0
  Metabolism and nutrition disorders: Severe | 0 | 0 | 0
  Musculoskeletal and connective disorders : Mild | 2 | 1 | 0
  Musculoskeletal and connective disorders : Moderate | 0 | 4 | 0
  Musculoskeletal and connective disorders : Severe | 1 | 3 | 0
  Nervous system disorders : Mild | 2 | 3 | 2
  Nervous system disorders : Moderate | 3 | 3 | 0
  Nervous system disorders : Severe | 2 | 2 | 0
  Psychiatric disorders: Mild | 2 | 0 | 0
  Psychiatric disorders: Moderate | 1 | 0 | 0
  Psychiatric disorders: Severe | 0 | 0 | 0
  Renal and urinary disorders: Mild | 1 | 0 | 0
  Renal and urinary disorders: Moderate | 0 | 0 | 0
  Renal and urinary disorders: Severe | 0 | 0 | 0
  Reproductive system and breast disorders : Mild | 0 | 1 | 0
  Reproductive system and breast disorders : Moderate | 0 | 1 | 0
  Reproductive system and breast disorders : Severe | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders : Mild | 4 | 1 | 1
  Respiratory, thoracic and mediastinal disorders : Moderate | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders : Severe | 0 | 0 | 0
  Skin and cutaneous tissue disorders : Mild | 3 | 7 | 1
  Skin and cutaneous tissue disorders : Moderate | 0 | 2 | 0
  Skin and cutaneous tissue disorders : Severe | 1 | 0 | 0

32. Primary Outcome: Frequency and Severity of Unsolicited Adverse Events by Treatment Group for Baseline ZIKV Seropositive and DENV Seropositive Participants
Description: as for outcome 29
Time Frame: Day 1 through Day 57
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Any SOC: Mild | 0 | 0 | 0
  Any SOC: Moderate | 1 | 0 | 0
  Any SOC: Severe | 0 | 0 | 0
  Infections and infestations: Mild | 0 | 0 | 0
  Infections and infestations: Moderate | 1 | 0 | 0
  Infections and infestations: Severe | 0 | 0 | 0

33. Primary Outcome: Frequency and Severity of Unsolicited Adverse Events by Treatment Group for Baseline ZIKV Seropositive and DENV Seronegative Participants
Description: Adverse events (AEs) are defined as any untoward medical occurrence regardless of its causal relationship to study treatment. Number of participants with an AE are summarized by MedDRA System Organ Class (SOC). Each participant was counted once per SOC. If a condition was present at screening, it was not considered an AE unless the severity worsened.
Time Frame: Day 1 through Day 57
Population: The Safety Analysis population includes all baseline ZIKV seropositvie and DENV seronegative participants who received at least one study vaccination. No subjects met the baseline ZIKV seropositive and DENV seronegative criteria.
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

34. Primary Outcome: Frequency and Severity of Unsolicited Adverse Events by Treatment Group for Baseline ZIKV Seronegative and DENV Seropositive Participants
Description: as for outcome 29
Time Frame: Day 1 through Day 57
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 26 | 33 | 9
Participants
  Any SOC : Mild | 16 | 21 | 4
  Any SOC : Moderate | 4 | 9 | 0
  Any SOC : Severe | 1 | 3 | 1
  Cardiac disorders : Mild | 0 | 2 | 0
  Cardiac disorders : Moderate | 0 | 0 | 0
  Cardiac disorders : Severe | 0 | 0 | 0
  Eye disorders : Mild | 0 | 2 | 0
  Eye disorders : Moderate | 1 | 1 | 0
  Eye disorders : Severe | 0 | 1 | 0
  Gastrointestinal disorders : Mild | 3 | 1 | 0
  Gastrointestinal disorders : Moderate | 0 | 1 | 0
  Gastrointestinal disorders : Severe | 0 | 0 | 0
  General disorders and administration site conditions : Mild | 2 | 2 | 1
  General disorders and administration site conditions : Moderate | 1 | 3 | 0
  General disorders and administration site conditions : Severe | 0 | 1 | 0
  Infections and infestations : Mild | 8 | 7 | 2
  Infections and infestations : Moderate | 1 | 2 | 0
  Infections and infestations : Severe | 0 | 3 | 0
  Injury, poisoning and procedural complications : Mild | 0 | 3 | 0
  Injury, poisoning and procedural complications : Moderate | 1 | 0 | 0
  Injury, poisoning and procedural complications : Severe | 0 | 0 | 1
  Investigations : Mild | 2 | 3 | 0
  Investigations : Moderate | 0 | 0 | 0
  Investigations : Severe | 0 | 0 | 0
  Metabolism and nutrition disorders : Mild | 1 | 0 | 0
  Metabolism and nutrition disorders : Moderate | 0 | 0 | 0
  Metabolism and nutrition disorders : Severe | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders : Mild | 1 | 1 | 0
  Musculoskeletal and connective tissue disorders : Moderate | 0 | 4 | 0
  Musculoskeletal and connective tissue disorders : Severe | 0 | 2 | 0
  Nervous system disorders : Mild | 2 | 3 | 2
  Nervous system disorders : Moderate | 2 | 3 | 0
  Nervous system disorders : Severe | 1 | 1 | 0
  Psychiatric disorders : Mild | 1 | 0 | 0
  Psychiatric disorders : Moderate | 1 | 0 | 0
  Psychiatric disorders : Severe | 0 | 0 | 0
  Renal and urinary disorders : Mild | 1 | 0 | 0
  Renal and urinary disorders : Moderate | 0 | 0 | 0
  Renal and urinary disorders : Severe | 0 | 0 | 0
  Reproductive system and breast disorders : Mild | 0 | 1 | 0
  Reproductive system and breast disorders : Moderate | 0 | 1 | 0
  Reproductive system and breast disorders : Severe | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders : Mild | 2 | 1 | 1
  Respiratory, thoracic and mediastinal disorders : Moderate | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders : Severe | 0 | 0 | 0
  Skin and subcutaneous tissue disorders : Mild | 3 | 6 | 1
  Skin and subcutaneous tissue disorders : Moderate | 0 | 2 | 0
  Skin and subcutaneous tissue disorders : Severe | 1 | 0 | 0

35. Primary Outcome: Frequency and Severity of Unsolicited Adverse Events by Treatment Group for Baseline ZIKV Seronegative and DENV Seronegative Participants
Description: as for outcome 29
Time Frame: Day 1 through Day 57
Population: The Safety Analysis population includes all participants baseline ZIKV seronegative and DENV seronegative participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 8 | 10 | 1
Participants
  Any SOC : Mild | 5 | 5 | 1
  Any SOC : Moderate | 1 | 2 | 0
  Any SOC : Severe | 1 | 1 | 0
  Eye disorders : Mild | 1 | 0 | 0
  Eye disorders : Moderate | 0 | 0 | 0
  Eye disorders : Severe | 0 | 0 | 0
  Cardiac disorders : Mild | 0 | 1 | 0
  Cardiac disorders : Moderate | 0 | 1 | 0
  Cardiac disorders : Severe | 0 | 0 | 0
  Gastrointestinal disorders : Mild | 1 | 0 | 0
  Gastrointestinal disorders : Moderate | 0 | 0 | 0
  Gastrointestinal disorders : Severe | 0 | 1 | 0
  General disorders and administration site conditions : Mild | 0 | 0 | 0
  General disorders and administration site conditions : Moderate | 0 | 0 | 0
  General disorders and administration site conditions : Severe | 1 | 1 | 0
  Immune system disorders : Mild | 0 | 0 | 0
  Immune system disorders : Moderate | 0 | 1 | 0
  Immune system disorders : Severe | 0 | 0 | 0
  Infections and infestations : Mild | 1 | 1 | 1
  Infections and infestations : Moderate | 0 | 0 | 0
  Infections and infestations : Severe | 0 | 1 | 0
  Injury, poisoning and procedural complications : Mild | 1 | 1 | 0
  Injury, poisoning and procedural complications : Moderate | 0 | 1 | 0
  Injury, poisoning and procedural complications : Severe | 0 | 0 | 0
  Investigations : Mild | 2 | 1 | 0
  Investigations : Moderate | 0 | 0 | 0
  Investigations : Severe | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders : Mild | 1 | 0 | 0
  Musculoskeletal and connective tissue disorders : Moderate | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders : Severe | 1 | 1 | 0
  Nervous system disorders : Mild | 0 | 0 | 0
  Nervous system disorders : Moderate | 1 | 0 | 0
  Nervous system disorders : Severe | 1 | 1 | 0
  Psychiatric disorders : Mild | 1 | 0 | 0
  Psychiatric disorders : Moderate | 0 | 0 | 0
  Psychiatric disorders : Severe | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders : Mild | 2 | 0 | 0
  Respiratory, thoracic and mediastinal disorders : Moderate | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders : Severe | 0 | 0 | 0
  Skin and subcutaneous tissue disorders : Mild | 0 | 1 | 0
  Skin and subcutaneous tissue disorders : Moderate | 0 | 0 | 0
  Skin and subcutaneous tissue disorders : Severe | 0 | 0 | 0

36. Primary Outcome: Frequency and Type of Serious Adverse Events (SAE) Considered Related to Study Vaccine for All Participants
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 750
Population: The Safety Analysis population includes all with available results who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 35 | 45 | 10
Participants | 0 | 0 | 0

37. Primary Outcome: Duration of Serious Adverse Events (SAE) Considered Related to Study Vaccine for All Participants
Description: as for outcome 36
Time Frame: Day 1 through Day 750
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 35 | 45 | 10
Participants | 0 | 0 | 0

38. Primary Outcome: Frequency and Type of Adverse Events of Special Interest (AESI) Considered Related to Study Vaccine for All Participants
Description: For this study Neurologic and Neuroinflammatory Disorders after the first vaccination were considered as Adverse Events of Special Interest (AESI).
Time Frame: Day 1 through Day 750
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 35 | 45 | 10
Participants | 0 | 0 | 0

39. Primary Outcome: Duration of Adverse Events of Special Interest (AESI) Considered Related to Study Vaccine for All Participants
Description: as for outcome 38
Time Frame: Day 1 through Day 750
Population: The Safety Analysis population includes all participants with available results who received at least one study vaccination. No AESIs were reported.
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

40. Primary Outcome: Frequency of New Onset Chronic Medical Conditions for All Participants
Description: New onset chronic medical conditions (NOCMCs) were any new medical conditions reported from the first administration of study vaccine until the end of the study.
Time Frame: Day 1 through Day 750
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 35 | 45 | 10
Participants
  All Participants | 1 | 0 | 0
  Baseline ZIKV Seropositive: number analyzed (Participants) | 1 | 1 | 0
  Baseline ZIKV Seropositive | 0 | 0 | 0
  Baseline ZIKV Seronegative: number analyzed (Participants) | 34 | 43 | 10
  Baseline ZIKV Seronegative | 1 | 0 | 0
  Baseline ZIKV Seropositive and DENV Seropositive: number analyzed (Participants) | 1 | 1 | 0
  Baseline ZIKV Seropositive and DENV Seropositive | 0 | 0 | 0
  Baseline Seropositive and DENV Seronegative: number analyzed (Participants) | 0 | 0 | 0
  Baseline Seropositive and DENV Seronegative | 0 | 0 | 0
  Baseline ZIKV Seronegative and DENV Seropositive: number analyzed (Participants) | 26 | 33 | 9
  Baseline ZIKV Seronegative and DENV Seropositive | 1 | 0 | 0
  Baseline ZIKV Seronegative and DENV Seronegative: number analyzed (Participants) | 8 | 10 | 1
  Baseline ZIKV Seronegative and DENV Seronegative | 0 | 0 | 0

41. Primary Outcome: Comparison of Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for All Participants
Description: The number of participants experiencing each adverse event are listed.
Time Frame: Day 1 through Day 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 35 | 45 | 10
Participants
  Vaccine-related Grade 3 local, systemic, or laboratory: Any Event | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 4 | 4 | 1
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Fever | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Headache | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Pain | 2 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness | 1 | 1 | 0

42. Primary Outcome: Comparison of the Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for All Participants
Description: The number of participants experiencing each adverse event are listed.
Time Frame: Day 29 through Day 36
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 32 | 43 | 9
Participants
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 1 | 5 | 0
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Fever | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Headache | 0 | 1 | 0
  Myalgia (Body Aches/Muscular Pain) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Pain | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Abdominal Pain | 1 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Malaise (General Unwell Feeling) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Nausea | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Vomiting | 0 | 1 | 0

43. Primary Outcome: Comparison of the Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for Baseline ZIKV Seropositive Participants
Description: The number of participants experiencing each adverse event are listed.
Time Frame: Day 1 through Day 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV
Number analyzed (Participants) | 1 | 1
Participants
  Vaccine related Grade 3 local, systemic or laboratory AE | 0 | 0
  Grade 2 or greater local or systemic reactogenicity | 0 | 0

44. Primary Outcome: Comparison of the Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for Baseline ZIKV Seropositive Participants
Description: The number of participants experiencing each adverse event are listed.
Time Frame: Day 29 through Day 36
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV
Number analyzed (Participants) | 1 | 1
Participants
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 0 | 0

45. Primary Outcome: Comparison of the Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for Baseline ZIKV Seronegative Participants
Description: The number of participants experiencing each adverse event are listed.
Time Frame: Day 1 through Day 8
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 34 | 43 | 10
Participants
  Vaccine related Grade 3 local, systemic or laboratory: Any Event | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 4 | 3 | 1
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Fever | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Headache | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) | 1 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Pain | 2 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness | 1 | 1 | 0

46. Primary Outcome: Comparison of the Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for Baseline ZIKV Seronegative Participants
Description: The number of participants experiencing each adverse event are listed.
Time Frame: Day 29 through Day 36
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 31 | 41 | 9
Participants
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 1 | 5 | 0
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Fever | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Headache | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Pain | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Abdominal Pain | 1 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Malaise (General Unwell Feeling) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Nausea | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Vomiting | 0 | 1 | 0

47. Primary Outcome: Comparison of the Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for Baseline ZIKV Seropositive and DENV Seropositive Participants
Description: The number of participants experiencing each adverse event are listed.
Time Frame: Day 1 through Day 8
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV
Number analyzed (Participants) | 1 | 1
Participants
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 0 | 0

48. Primary Outcome: Comparison of the Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for Baseline ZIKV Seropositive and DENV Seropositive Participants
Description: The number of participants experiencing each adverse event are listed.
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all baseline ZIKV positive and DENV seropositive participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV
Number analyzed (Participants) | 1 | 1
Participants
  Vaccine related Grade 3 local, systemic, or laboratory AE: Any Event | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 0 | 0

49. Primary Outcome: Comparison of the Frequency, Type, and Duration of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for Baseline ZIKV Seropositive and DENV Seronegative Participants
Description: The number of participants experiencing each adverse event and the median duration of adverse events are listed.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seropositive and DENV seronegative participants who received at least one study vaccination. No participants met the baseline ZIKV seropositive and DENV seronegative criteria.
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

50. Primary Outcome: Comparison of the Frequency, Type, and Duration of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for Baseline ZIKV Seropositive and DENV Seronegative Participants
Description: The number of participants experiencing each adverse event and the median duration of adverse events are listed.
Time Frame: Day 29 through Day 36
Population: as for outcome 49
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

51. Primary Outcome: Comparison of the Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for Baseline ZIKV Seronegative and DENV Seropositive Participants
Description: The number of participants experiencing each adverse event are listed.
Time Frame: Day 1 through Day 8
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 26 | 33 | 9
Participants
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 3 | 3 | 1
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) | 0 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Fever | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Headache | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) | 1 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Pain | 2 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness | 1 | 1 | 0

52. Primary Outcome: Comparison of the Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for Baseline ZIKV Seronegative and DENV Seropositive Participants
Description: The number of participants experiencing each adverse event will be listed
Time Frame: Day 29 through Day 36
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 23 | 31 | 8
Participants
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 1 | 4 | 0
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Pain | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Abdominal Pain | 1 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Malaise (General Unwell Feeling) | 0 | 1 | 0

53. Primary Outcome: Comparison of the Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for Baseline ZIKV Seronegative and DENV Seronegative Participants
Description: The number of participants experiencing each adverse event are listed.
Time Frame: Day 1 through Day 8
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 8 | 10 | 1
Participants
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 1 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) | 1 | 0 | 0

54. Primary Outcome: Comparison of the Frequency and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for Baseline ZIKV Seronegative and DENV Seronegative Participants
Description: The number of participants experiencing each adverse event are listed.
Time Frame: Day 29 through Day 36
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 8 | 10 | 1
Participants
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Fever | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Headache | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Abdominal Pain | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Malaise (General Unwell Feeling) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Nausea | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Vomiting | 0 | 1 | 0

55. Primary Outcome: Comparison of the Duration and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for All Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants with available results who received at least one study vaccination and experienced an event as reported in Outcome Measure 41.
Measure: Median (Full Range); unit: Days
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 4 | 4 | 1
Days
  Vaccine-related Grade 3 local, systemic, or laboratory: Any Event: number analyzed (Participants) | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 2.5 [1 to 7] | 2 [1 to 4] | 1.5 [1 to 3]
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain): number analyzed (Participants) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) |  |  | 1 [1 to 1]
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness): number analyzed (Participants) | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) | 4 [4 to 4] | 1 [1 to 1] | 3 [3 to 3]
  Grade 2 or greater local or systemic reactogenicity: Fever: number analyzed (Participants) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Fever |  |  | 2 [2 to 2]
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating): number analyzed (Participants) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) |  |  | 1 [1 to 1]
  Grade 2 or greater local or systemic reactogenicity: Headache: number analyzed (Participants) | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Headache | 7 [7 to 7] | 4 [4 to 4] | 3 [3 to 3]
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain): number analyzed (Participants) | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) | 3 [3 to 3] | 2 [2 to 2] | 1 [1 to 1]
  Grade 2 or greater local or systemic reactogenicity: Pain: number analyzed (Participants) | 2 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Pain | 1.5 [1 to 2] | 2 [2 to 2] |
  Grade 2 or greater local or systemic reactogenicity: Tenderness: number analyzed (Participants) | 1 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness | 2 [2 to 2] | 2 [2 to 2] |

56. Primary Outcome: Comparison of the Duration and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for All Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all participants with available results who received at least one study vaccination and experienced an event as reported in Outcome Measure 42.
Measure: Median (Full Range); unit: Days
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 5 | 0
Days
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event: number analyzed (Participants) | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 1 [1 to 1] | 2 [1 to 11] |
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain): number analyzed (Participants) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) |  | 5.5 [1 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness): number analyzed (Participants) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) |  | 7.5 [4 to 11] |
  Grade 2 or greater local or systemic reactogenicity: Fever: number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Fever |  | 1 [1 to 1] |
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating): number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) |  | 3 [3 to 3] |
  Grade 2 or greater local or systemic reactogenicity: Headache: number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Headache |  | 10 [10 to 10] |
  Myalgia (Body Aches/Muscular Pain): number analyzed (Participants) | 0 | 2 | 0
  Myalgia (Body Aches/Muscular Pain) |  | 5.5 [1 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Pain: number analyzed (Participants) | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Pain |  | 2 [1 to 2] |
  Grade 2 or greater local or systemic reactogenicity: Tenderness: number analyzed (Participants) | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness |  | 2 [1 to 2] |
  Grade 2 or greater local or systemic reactogenicity: Abdominal Pain: number analyzed (Participants) | 1 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Abdominal Pain | 1 [1 to 1] | 1 [1 to 1] |
  Grade 2 or greater local or systemic reactogenicity: Malaise (General Unwell Feeling): number analyzed (Participants) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Malaise (General Unwell Feeling) |  | 7.5 [5 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Nausea: number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Nausea |  | 3 [3 to 3] |
  Grade 2 or greater local or systemic reactogenicity: Vomiting: number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Vomiting |  | 1 [1 to 1] |

57. Primary Outcome: Comparison of the Duration and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for Baseline ZIKV Seropositive Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seropositive participants who received at least one study vaccination and experienced an event as reported in Outcome Measure 43.
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

58. Primary Outcome: Comparison of the Duration and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for Baseline ZIKV Seropositive Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all baseline ZIKV seropositive participants who received at least one study vaccination and experienced an event as reported in Outcome Measure 44.
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

59. Primary Outcome: Comparison of the Duration and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for Baseline ZIKV Seronegative Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seronegative participants who received at least one study vaccination and experienced an event as reported in Outcome Measure 45.
Measure: Median (Full Range); unit: Days
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 4 | 3 | 1
Days
  Vaccine related Grade 3 local, systemic or laboratory: Any Event: number analyzed (Participants) | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 2.5 [1 to 7] | 2 [1 to 4] | 1.5 [1 to 3]
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain): number analyzed (Participants) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) |  |  | 1 [1 to 1]
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness): number analyzed (Participants) | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) | 4 [4 to 4] | 1 [1 to 1] | 3 [3 to 3]
  Grade 2 or greater local or systemic reactogenicity: Fever: number analyzed (Participants) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Fever |  |  | 2 [2 to 2]
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating): number analyzed (Participants) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) |  |  | 1 [1 to 1]
  Grade 2 or greater local or systemic reactogenicity: Headache: number analyzed (Participants) | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Headache | 7 [7 to 7] | 4 [4 to 4] | 3 [3 to 3]
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain): number analyzed (Participants) | 1 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) | 3 [3 to 3] |  | 1 [1 to 1]
  Grade 2 or greater local or systemic reactogenicity: Pain: number analyzed (Participants) | 2 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Pain | 1.5 [1 to 2] | 2 [2 to 2] |
  Grade 2 or greater local or systemic reactogenicity: Tenderness: number analyzed (Participants) | 1 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness | 2 [2 to 2] | 2 [2 to 2] |

60. Primary Outcome: Comparison of the Duration and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for Baseline ZIKV Seronegative Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all baseline ZIKV seronegative participants who received at least one study vaccination and experienced an event as reported in Outcome Measure 46.
Measure: Median (Full Range); unit: Days
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 5 | 0
Days
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event: number analyzed (Participants) | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 1 [1 to 1] | 2 [1 to 11] |
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain): number analyzed (Participants) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) |  | 5.5 [1 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness): number analyzed (Participants) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) |  | 7.5 [4 to 11] |
  Grade 2 or greater local or systemic reactogenicity: Fever: number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Fever |  | 1 [1 to 1] |
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating): number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) |  | 3 [3 to 3] |
  Grade 2 or greater local or systemic reactogenicity: Headache: number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Headache |  | 10 [10 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain): number analyzed (Participants) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) |  | 5.5 [1 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Pain: number analyzed (Participants) | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Pain |  | 2 [1 to 2] |
  Grade 2 or greater local or systemic reactogenicity: Tenderness: number analyzed (Participants) | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness |  | 2 [1 to 2] |
  Grade 2 or greater local or systemic reactogenicity: Abdominal Pain: number analyzed (Participants) | 1 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Abdominal Pain | 1 [1 to 1] | 1 [1 to 1] |
  Grade 2 or greater local or systemic reactogenicity: Malaise (General Unwell Feeling): number analyzed (Participants) | 0 | 2 | 0
  Grade 2 or greater local or systemic reactogenicity: Malaise (General Unwell Feeling) |  | 7.5 [5 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Nausea: number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Nausea |  | 3 [3 to 3] |
  Grade 2 or greater local or systemic reactogenicity: Vomiting: number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Vomiting |  | 1 [1 to 1] |

61. Primary Outcome: Comparison of the Duration and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for Baseline ZIKV Seropositive and DENV Seropositive Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seropositive and DENV seropositive participants who received at least one study vaccination and experienced an event as reported in Outcome Measure 47.
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

62. Primary Outcome: Comparison of the Duration and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for Baseline ZIKV Seropositive and DENV Seropositive Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all baseline ZIKV positive and DENV seropositive participants who received at least one study vaccination and experienced an event as reported in Outcome Measure 48.
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

63. Primary Outcome: Comparison of the Duration and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for Baseline ZIKV Seronegative and DENV Seropositive Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seronegative and DENV seropositive participants who received at least one study vaccination and experienced an event as reported in Outcome Measure 51.
Measure: Median (Full Range); unit: Days
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 3 | 3 | 1
Days
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event: number analyzed (Participants) | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 2 [1 to 7] | 2 [1 to 4] | 1.5 [1 to 3]
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain): number analyzed (Participants) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) |  |  | 1 [1 to 1]
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness): number analyzed (Participants) | 0 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) |  | 1 [1 to 1] | 3 [3 to 3]
  Grade 2 or greater local or systemic reactogenicity: Fever: number analyzed (Participants) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Fever |  |  | 2 [2 to 2]
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating): number analyzed (Participants) | 0 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) |  |  | 1 [1 to 1]
  Grade 2 or greater local or systemic reactogenicity: Headache: number analyzed (Participants) | 1 | 1 | 1
  Grade 2 or greater local or systemic reactogenicity: Headache | 7 [7 to 7] | 4 [4 to 4] | 3 [3 to 3]
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain): number analyzed (Participants) | 1 | 0 | 1
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) | 3 [3 to 3] |  | 1 [1 to 1]
  Grade 2 or greater local or systemic reactogenicity: Pain: number analyzed (Participants) | 2 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Pain | 1.5 [1 to 2] | 2 [2 to 2] |
  Grade 2 or greater local or systemic reactogenicity: Tenderness: number analyzed (Participants) | 1 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness | 2 [2 to 2] | 2 [2 to 2] |

64. Primary Outcome: Comparison of the Duration and Type Duration of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for Baseline ZIKV Seronegative and DENV Seropositive Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all baseline ZIKV seronegative and DENV seropositive participants who received at least one study vaccination and experienced an event as reported in Outcome Measure 52.
Measure: Median (Full Range); unit: Days
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 4 | 0
Days
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event: number analyzed (Participants) | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 1 [1 to 1] | 2 [1 to 11] |
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain): number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) |  | 1 [1 to 1] |
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness): number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) |  | 11 [11 to 11] |
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain): number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) |  | 1 [1 to 1] |
  Grade 2 or greater local or systemic reactogenicity: Pain: number analyzed (Participants) | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Pain |  | 2 [1 to 2] |
  Grade 2 or greater local or systemic reactogenicity: Tenderness: number analyzed (Participants) | 0 | 3 | 0
  Grade 2 or greater local or systemic reactogenicity: Tenderness |  | 2 [1 to 2] |
  Grade 2 or greater local or systemic reactogenicity: Abdominal Pain: number analyzed (Participants) | 1 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Abdominal Pain | 1 [1 to 1] |  |
  Grade 2 or greater local or systemic reactogenicity: Malaise (General Unwell Feeling): number analyzed (Participants) | 0 | 1 | 0
  Grade 2 or greater local or systemic reactogenicity: Malaise (General Unwell Feeling) |  | 5 [5 to 5] |

65. Primary Outcome: Comparison of the Duration and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 1 for Baseline ZIKV Seronegative and DENV Seronegative Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all baseline ZIKV seronegative and DENV seronegative participants who received at least one study vaccination and experienced an event as reported in Outcome Measure 53.
Measure: Median (Full Range); unit: Days
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 0 | 0
Days
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event: number analyzed (Participants) | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event | 4 [4 to 4] |  |
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) | 4 [4 to 4] |  |

66. Primary Outcome: Comparison of the Duration and Type of Vaccine-related Grade 3 Local, Systemic, or Laboratory AE, and Grade 2 or Greater Local or Systemic Reactogenicity Post Dose 2 for Baseline ZIKV Seronegative and DENV Seronegative Participants
Description: The median duration of adverse events are listed.
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all baseline ZIKV seronegative and DENV seronegative participants who received at least one study vaccination and experienced an event as reported in Outcome Measure 54.
Measure: Median (Full Range); unit: Days
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 1 | 0
Days
  Vaccine related Grade 3 local, systemic or laboratory AE: Any Event: number analyzed (Participants) | 0 | 0 | 0
  Grade 2 or greater local or systemic reactogenicity: Any Event |  | 3.5 [1 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Arthralgia (Joint Pain) |  | 10 [10 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Fatigue (Tiredness) |  | 4 [4 to 4] |
  Grade 2 or greater local or systemic reactogenicity: Fever |  | 1 [1 to 1] |
  Grade 2 or greater local or systemic reactogenicity: Feverishness (Chills/Shivering/Sweating) |  | 3 [3 to 3] |
  Grade 2 or greater local or systemic reactogenicity: Headache |  | 10 [10 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Myalgia (Body Aches/Muscular Pain) |  | 10 [10 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Abdominal Pain |  | 1 [1 to 1] |
  Grade 2 or greater local or systemic reactogenicity: Malaise (General Unwell Feeling) |  | 10 [10 to 10] |
  Grade 2 or greater local or systemic reactogenicity: Nausea |  | 3 [3 to 3] |
  Grade 2 or greater local or systemic reactogenicity: Vomiting |  | 1 [1 to 1] |

67. Primary Outcome: Comparison of Study Withdrawals and Discontinuation of Study Vaccination Due to Any Reason for All Participants
Description: Comparisons of the number of participants who withdrew early and who discontinued treatment are presented.
Time Frame: Day 1 through Day 750
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 36 | 45 | 10
Participants
  Withdrew from Study | 10 | 13 | 4
  Discontinuation of Study Vaccination | 3 | 2 | 1

68. Primary Outcome: Comparison of Study Withdrawals and Discontinuation of Study Vaccination Due to Any Reason for Baseline ZIKV Seropositive Participants
Description: Comparisons of the number of participants who withdrew early and who discontinued treatment are presented.
Time Frame: Day 1 through Day 750
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Withdrew from Study | 0 | 1 | 0
  Discontinuation of Study Vaccination | 0 | 0 | 0

69. Primary Outcome: Comparison of Study Withdrawals and Discontinuation of Study Vaccination Due to Any Reason for Baseline ZIKV Seronegative Participants
Description: Comparisons of the number of participants who withdrew early and who discontinued treatment are presented.
Time Frame: Day 1 through Day 750
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 34 | 43 | 10
Participants
  Withdrew from Study | 9 | 12 | 4
  Discontinuation of Study Vaccination | 3 | 2 | 1

70. Primary Outcome: Comparison of Study Withdrawals and Discontinuation of Study Vaccination Due to Any Reason for Baseline ZIKV Seropositive and DENV Seropositive Participants
Description: Comparisons of the number of participants who withdrew early and who discontinued treatment are presented.
Time Frame: Day 1 through Day 750
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 1 | 1 | 0
Participants
  Withdrew from Study | 0 | 1 | 0
  Discontinuation of Study Vaccination | 0 | 0 | 0

71. Primary Outcome: Comparison of Study Withdrawals and Discontinuation of Study Vaccination Due to Any Reason for Baseline ZIKV Seropositive and DENV Seronegative Participants
Description: Comparisons of the number of participants who withdrew early and who discontinued treatment are presented.
Time Frame: Day 1 through Day 750
Population: as for outcome 23
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 0 | 0 | 0

72. Primary Outcome: Comparison of Study Withdrawals and Discontinuation of Study Vaccination Due to Any Reason for Baseline ZIKV Seronegative and DENV Seropositive Participants
Description: Comparisons of the number of participants who withdrew early and who discontinued treatment are presented.
Time Frame: Day 1 through Day 750
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 26 | 33 | 9
Participants
  Withdrew from Study | 7 | 10 | 4
  Discontinuation of Study Vaccination | 3 | 2 | 1

73. Primary Outcome: Comparison of Study Withdrawals and Discontinuation of Study Vaccination Due to Any Reason for Baseline ZIKV Seronegative and DENV Seronegative Participants
Description: Comparisons of the number of participants who withdrew early and who discontinued treatment are presented.
Time Frame: Day 1 through Day 750
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
Number analyzed (Participants) | 8 | 10 | 1
Participants
  Withdrew from Study | 2 | 2 | 0
  Discontinuation of Study Vaccination | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited Adverse Events (AEs) were collected from the time of each study vaccination through 8 days post-vaccination and unsolicited AEs were collected from the time of first study vaccination through 28 days after last study vaccination. New-onset chronic medical conditions, Serious AEs and Adverse Events of Special Interest (AESIs) were collected from the time of first study vaccination through end of study follow up period (approximately 24 months).
Description: Solicited AEs included local reactions and systemic reactions. Local (injection site) reactions included pain, tenderness, pruritus, ecchymosis, erythema, and induration/swelling. Systemic reactions included fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, nausea, vomiting, diarrhea, abdominal pain, and rash.
Arm/Group | 2.5 mcg ZPIV | 5 mcg ZPIV | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/45 | 1/10
Serious Adverse Events (participants affected / at risk) | 2/35 | 1/45 | 1/10
Other Adverse Events (participants affected / at risk) | 20/35 | 29/45 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5 mcg ZPIV (N=35) | 5 mcg ZPIV (N=45) | Placebo (N=10)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Schizoaffective disorder bipolar type (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5 mcg ZPIV (N=35) | 5 mcg ZPIV (N=45) | Placebo (N=10)
Bradycardia (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
Eye pain (Eye disorders) | 2 (2) | 3 (3) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 4 (4) | 5 (5) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 5 (5) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 2 (2) | 3 (4) | 0 (0)
Blood pressure systolic decreased (Investigations) | 3 (4) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 7 (8) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (6) | 7 (17) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT03008122/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT03008122/SAP_001.pdf